CLINICAL TRIAL: NCT06332768
Title: Comparison of High Flow Oxygenation, Noninvasive Ventilation and Standard Oxygen Therapy in the Early Post-extubation Period in Patients With Acute Respiratory Distress Syndrome
Brief Title: NIV Versus HFO Versus Standard Therapy Immediately After Weaning From Mechanical Ventilation in ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Principal Investigator, Mikhail Y. Kirov, Head of the anesthesiology and intensive care department, Northern State Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: WEAN_2021
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Mechanical Ventilation Complication; Weaning Failure; Acute Respiratory Distress Syndrome; High-flow Oxygenation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIV (Active Comparator): Non-invasive ventilation
  Interventions: Device: Respiratory support
- HFO (Active Comparator): High Flow Oxygenation
  Interventions: Device: Respiratory support

INTERVENTIONS:
Device: Respiratory support — High-flow nasal oxygenation
  Other Names: Oxygenation

SUMMARY:
The weaning failure is a paramount challenge when aggressive discontinuation of respiratory support in ARDS. The aim of the study is to improve weaning safety and efficacy by a transient postextubation non-invasive respiratory support.

DETAILED DESCRIPTION:
HFNO (high-flow nasal oxygenation and NIV (non invasive ventilation) are to be randomly compared in the ARDS postextubation period.

ELIGIBILITY:
Inclusion Criteria:

ARDS

Exclusion Criteria:

Severe ICU-aquired weakness Severe COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Weaning failure | 48 hrs
  Weaning failure and re-intubation or recanulation

CONTACTS AND LOCATIONS:
Locations (1):
- City hospital # 1, Arkhangelsk, Arkhangelskaya oblast, Russia